CLINICAL TRIAL: NCT00001761
Title: Phase I Trial of Recombinant Human Interleukin-10 (SCH 52000) in Patients With Wegener's Granulomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980059; 98-I-0059
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-01

CONDITIONS: Vasculitis; Wegener's Granulomatosis
Keywords: Autoimmunity; Cytokine; Inflammation; Interleukin; Vasculitis; Wegener's Granulomatosis
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis; Autoimmune Diseases; Inflammation | interventions — Interleukin-10

INTERVENTIONS:
Drug: Interleukin-10

SUMMARY:
The purpose of this study is to assess the safety, tolerance, and immunologic effects of interleukin-10 (IL-10), in patients with Wegener's granulomatosis. A secondary objective is to determine if IL-10 demonstrates sufficient anti-inflammatory activity in the treatment of Wegener's granulomatosis to warrant further study in a larger trial. In this study, IL-10 will be given either alone or in combination with standard therapeutic agents, usually consisting of cyclophosphamide, methotrexate, and/or prednisone. Patients will be eligible to receive IL-10 when there is evidence of active disease. IL-10 will be administered by subcutaneous injection at a dose of 4 µ (Micro)g/kg/day for 28 days.

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety, tolerance, and immunologic effects of interleukin-10 (IL-10), in patients with Wegener's granulomatosis. A secondary objective is to determine if IL-10 demonstrates sufficient anti-inflammatory activity in the treatment of Wegener's granulomatosis to warrant further study in a larger trial. In this study, IL-10 will be given either alone or in combination with standard therapeutic agents, usually consisting of cyclophosphamide, methotrexate, and/or prednisone. Patients will be eligible to receive IL-10 when there is evidence of active disease. IL-10 will be administered by subcutaneous injection at a dose of 4 µ (Micro)g/kg/day for 28 days.

ELIGIBILITY:
Diagnosis of Wegener's granulomatosis based on clinical characteristics and histopathological and/or angiographic evidence of vasculitis or the presence of glomerulonephritis and a positive assay for anti-neutrophil cytoplasmic autoantibodies (ANCA).

Age between 18 to 65 years.

No change in immunosuppressive drug therapy during the prior 4 weeks and one of the following:

Persistent disease activity ("Vasculitis Activity Index" score of greater than or equal to 3) despite optimal therapy;

Persistent or recurrent disease activity in a patient who cannot tolerate optimal therapy;

Patients not on maximal immunosuppressive therapy but with persistent or recurrent disease activity that is not, in the judgment of investigators, immediately threatening the function of a major organ system;

No evidence of active infection.

Patients may not be pregnant or nursing infants. Fertile women must have a negative pregnancy test within one week prior to study entry and all participants must be using effective means of birth control.

Serum creatinine is less than 3.5 mg/dL.

Hemocytopenia (platelet count is greater than 100,000/mm(3), leukocyte count is greater than 3,500/mm(s), hemoglobin is greater than 9 mg/dL).

Liver function test abnormalities is less than 3x upper limits of normal (either serum GOT, GPT, alkaline phosphatase, and/or bilirubin).

Patients cannot be anti-HIV, anti-HCV, or anti-Hepatitis B surface antigen (HBsAG) positive.

Weight greater less than 104 Kg (because of SCH 52000 concentration and volume limitations for subcutaneous injection).

No treatment with any investigational drug within 30 days.

No pre-existing malignancy.

No known allergy to E. coli protein or IL-10.

No history of psychiatric illness that in the opinion of the principal investigator would preclude entrance into the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 1998-02; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hoffman GS, Kerr GS, Leavitt RY, Hallahan CW, Lebovics RS, Travis WD, Rottem M, Fauci AS. Wegener granulomatosis: an analysis of 158 patients. Ann Intern Med. 1992 Mar 15;116(6):488-98. doi: 10.7326/0003-4819-116-6-488. PMID 1739240
- [Background] Ludviksson BR, Sneller MC, Chua KS, Talar-Williams C, Langford CA, Ehrhardt RO, Fauci AS, Strober W. Active Wegener's granulomatosis is associated with HLA-DR+ CD4+ T cells exhibiting an unbalanced Th1-type T cell cytokine pattern: reversal with IL-10. J Immunol. 1998 Apr 1;160(7):3602-9. PMID 9531324